CLINICAL TRIAL: NCT01831895
Title: CALM-FIM_US -Controlling and Lowering Blood Pressure With the MobiusHD™ - A Prospective Multicenter Safety Study
Brief Title: Controlling and Lowering Blood Pressure With The MOBIUSHD™
Acronym: CALM-FIM_US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Dynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALM-FIM_US, CRD0152, G130013
Record Dates: First submitted 2013-04-09; First posted 2013-04-15 (Estimated); Results first posted 2022-03-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: Hypertension; Carotid Sinus
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MobiusHD™ (Experimental): MobiusHD™
  Interventions: Device: MobiusHD™

INTERVENTIONS:
Device: MobiusHD™ — Implant that is placed in the carotid sinus to control hypertension.

SUMMARY:
To evaluate the safety and performance of the MobiusHD system in subjects with resistant hypertension.

DETAILED DESCRIPTION:
This is an open-label, multicenter, first-in-man clinical trial to be conducted inside the United States. Eligible subjects with stage 2 resistant systemic arterial hypertension currently being treated with a minimum of three (3) anti-hypertensive drugs, who consent to study participation will be assigned to treatment with the MobiusHD system.

Potential study participants will be consented and then screened at two (2) baseline visits beginning at least 30 days prior to MobiusHD placement. Qualified patients will undergo placement of the MobiusHD under angiographic visualization, and will then be followed for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Office cuff SBP ≥ 160 mmHg measured per protocol instructions (Appendix IV) following at least one (1) month of maximally tolerated therapy with at least three (3) anti-hypertensive medications, of which at least one (1) must be a diuretic. Any combination medications will be counted per the active ingredient. (For example, Zestoretic (Lisinopril +HCTZ) equals two (2) anti-hypertensive medications)

Exclusion Criteria:

* Known or clinically suspected baroreflex failure or autonomic neuropathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Bates, MD, Principal Investigator — West Virginia University
Locations (7):
- United States (7):
  - Cardiology, P.C., Birmingham, Alabama
  - Emory University, Atlanta, Georgia
  - Iowa Heart Center, Des Moines, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Rochester, Rochester, New York
  - The Carl & Edyth Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - Turkey Creek Medical Center, Knoxville, Tennessee

REFERENCES:
- [Derived] van Kleef MEAM, Devireddy CM, van der Heyden J, Bates MC, Bakris GL, Stone GW, Williams B, Spiering W; CALM-FIM Investigators. Treatment of Resistant Hypertension With Endovascular Baroreflex Amplification: 3-Year Results From the CALM-FIM Study. JACC Cardiovasc Interv. 2022 Feb 14;15(3):321-332. doi: 10.1016/j.jcin.2021.12.015. PMID 35144789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MobiusHD™
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | MobiusHD™
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 55.4 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Systolic Office Blood Pressure [Mean (Full Range); unit: mmHg] | 177 [160 to 203]

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of Participants with Adverse Events
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | MobiusHD™
Number analyzed (Participants) | 17
participants
  Hypotension - acute | 1
  Abnormal lab finding - hypokalemia | 1
  Access site complication - hemorrhage - groin | 1
  Access site complication - postprocedural | 1
  Anesthia complications - blurred vision | 1
  Digestive system disorder - nausea | 1
  Digestive system disorder - vomiting | 1
  Hypertension - acute | 1
  Pain - head | 1
  Pain - puncture site | 2
  Respiratory abnormalities - upper respiratory infection | 1

2. Secondary Outcome: Change in Systolic Office Blood Pressure (OBP)
Description: Change in Systolic Office Blood Pressure (OBP) compared to baseline.
Time Frame: 3 years
Population: Of the 17 subjects enrolled, 1 subject died and 1 subject withdrew from the study. The remaining 15 subjects completed all study visits through 3 years.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MobiusHD™
Number analyzed (Participants) | 17
mmHg
  Discharge | -26.6 (18.1)
  7 days | -19 (22.9)
  30 days | -18.8 (20.9)
  90 days: number analyzed (Participants) | 16
  90 days | -23.3 (25.8)
  180 days: number analyzed (Participants) | 16
  180 days | -27.5 (22.6)
  1 year: number analyzed (Participants) | 16
  1 year | -20.8 (28.7)
  1.5 years: number analyzed (Participants) | 15
  1.5 years | -19.7 (32.5)
  2 years: number analyzed (Participants) | 15
  2 years | -20.3 (35.4)
  2.5 years: number analyzed (Participants) | 15
  2.5 years | -11.3 (32.4)
  3 years: number analyzed (Participants) | 15
  3 years | -18.2 (37.1)

3. Secondary Outcome: Change in Systolic Ambulatory Blood Pressure (ABPM)
Description: Change in Systolic Ambulatory Blood Pressure (ABPM) measured at 3 and 6 months compared to baseline values.
Time Frame: 6 months
Population: Of the 17 subjects enrolled in the study, 16 subjects were available for for systolic ABPM measurements at 3 and 6 months.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MobiusHD™
Number analyzed (Participants) | 16
mmHg
  3 months | -11.94 (19.69)
  6 months | -16.00 (17.91)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion (3 years).
Arm/Group | MobiusHD™
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 7/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MobiusHD™ (N=17)
Hypotension - acute (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MobiusHD™ (N=17)
Pain - puncture site (Skin and subcutaneous tissue disorders) | 2 (2)
Abnormal lab finding - hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Access site complication - hemorrhage - groin (Skin and subcutaneous tissue disorders) | 1 (1)
Access site complications - postprocedural (Skin and subcutaneous tissue disorders) | 1 (1)
Anesthesia complications - blurred vision (Eye disorders) | 1 (1)
Arrhythmia - Bradycardia (Cardiac disorders) | 1 (1)
Digestive system disorder - nausea (Gastrointestinal disorders) | 1 (1)
Digestive system disorder - vomitting (Gastrointestinal disorders) | 1 (1)
Hypertension - acute (Cardiac disorders) | 1 (1)
Pain - head (General disorders) | 1 (1)
Respiratory Abnormalities - Upper Respiratory Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT01831895/Prot_SAP_000.pdf